CLINICAL TRIAL: NCT01612429
Title: Amino Acid Therapy to Modify Protein Carbamylation in End Stage Renal Disease
Brief Title: Carbamylation in Renal Disease-modulation With Amino Acid Therapy
Acronym: CarRAAT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ravi Thadhani, Director of Clinical Research in Nephrology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-P-000775; IRB# 12-303 (Other: NEIRB)
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: Carbamylation; Albumin; Protein structure; Kidney disease
MeSH Terms: conditions — Kidney Diseases | interventions — Amino Acids, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amino acid supplementation (Experimental): Up to 500 mL of 5.4% amino acid solution (NephrAmine) by intravenous infusion 3 x weekly for 6 weeks.
  Interventions: Dietary Supplement: Amino acid supplementation

INTERVENTIONS:
Dietary Supplement: Amino acid supplementation — Single arm study in which dialysis patients will receive up to 500 mL of NephrAmine® (5.4% amino acids for injection; B. Braun Medical, Inc) containing 26.8 grams of essential amino acids at 125 mL/h during each dialysis session (3 times weekly for 6 weeks)
  Other Names: NephrAmine®

SUMMARY:
This is a pilot study to evaluate the effects of amino acid supplementation on the structure of certain proteins in the blood of dialysis patients. Patients with end stage renal disease (ESRD) usually have high levels of urea that may interact with blood proteins and change their structure by a process known as carbamylation. The investigators are interested in determining whether carbamylation is linked to adverse outcomes in dialysis patients and have hypothesized that supplementation with a balanced formulation of amino acids can reduce the amount of carbamylation that occurs. In this study, dialysis patients (n= up to 30) will receive intravenous supplementation with an FDA-approved amino acid solution (NephrAmine®, 5.4% amino acids) during regular dialysis sessions (3 times weekly for 6 weeks). During the 6 weeks of therapy and for 2 weeks of follow-up, blood will be drawn from patients' existing hemodialysis access ports (~60 ml total per month) to measure levels of carbamylated albumin, amino acids, and standard laboratory values. Patients will be closely monitored for safety and tolerability of the amino acid therapy. For each treated subject, we will follow an additional individual that is not receiving treatment to serve as a control (no intervention).

DETAILED DESCRIPTION:
As human kidney function declines so does the ability to excrete urea, the chief end product of nitrogen metabolism. Though elevated blood urea levels denote a loss of kidney function, they may also serve as a source for the pathophysiological consequences of kidney failure. Urea spontaneously dissociates to form cyanate, which in its unprotonated form can react with protein amino groups in a process known as carbamylation. Carbamylation-induced protein alterations may be involved in the progression of various diseases by changing the structure, charge, and function of enzymes, hormones, receptors, and amino acids. For example, proteins as diverse as collagen and low density lipoproteins (LDLs), are shown to induce the characteristic biochemical events of atherosclerosis progression when carbamylated. Our research seeks to examine how protein carbamylation contributes to the pathological sequelae of end stage renal disease (ESRD) and determine if novel therapeutics can attenuate this process.

Percent carbamylated albumin level can be used as a measure of overall carbamylation burden. Our preliminary work shows a negative correlation between subjects' percent carbamylated albumin level and circulating amino acids, suggesting that free amino acids may be active scavengers for reactive isocyanate. Furthermore, ex vivo studies show that amino acid supplementation attenuates the carbamylation reaction from occurring. To better assess the biologic pathways affecting carbamylation in dialysis patients and to bring discoveries closer to clinical and therapeutic application, we aim to conduct a pilot study evaluating the effect of amino acid supplementation on carbamylation in participants with ESRD undergoing maintenance hemodialysis. We believe elevated urea and amino acid deficiencies may play dominant roles in the carbamylation of proteins in ESRD and protein carbamylation may be modifiable by amino acid therapy. The proposed pilot study will directly assess this concept.

The specific aims of the study are to evaluate the effect of amino acid supplementation on carbamylation in ESRD patients undergoing maintenance hemodialysis: (1) by evaluating safe and optimal amino acid supplement dosing and (2) by investigating the effect of amino acid supplementation on plasma carbamylated albumin levels.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the investigational nature of the study and sign written informed consent
* Willing and able to adhere to all study-related procedures, including adherence to study medication regimen
* ≥18 years old
* On stable medical therapy in the last 30 days before the study entry, defined as no change, addition, or removal of medications
* Patients must satisfy the following criteria based on the initial screening laboratory values:
* Serum albumin ≥ 3.0 g/dL (30 g/L)
* Dialysis adequacy recorded as Kt/ V > 1.2
* Women of childbearing potential must be practicing barrier or oral contraception, for the duration of the study-related treatment, or be documented as surgically sterile or one year post-menopausal
* If female, be non-nursing, non-pregnant and have a negative pregnancy test within two weeks of starting study treatment
* On stable hemodialysis therapy for at least 90 days before the study entry, defined as receiving thrice weekly dialysis and carrying a diagnosis of ESRD
* Prescribed a dialysis treatment time of 4 hours per session

Exclusion Criteria:

* Taking any type of amino acid supplementation within the last 90 days
* Received parenteral nutrition within last 90 days
* History of allergy to any amino acid compound
* Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg during any of the previous 3 dialysis sessions (confirmed by repeat)
* Severe hepatic impairment
* Condition with prognosis <1 year at time of study entry
* Current active treatment in another investigational study or participation in another investigational study in the 1 month prior to screening
* Active malignancies or other serious concurrent or recent medical or psychiatric condition which, in the opinion of the Investigator, makes the patient unsuitable for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in plasma carbamylated albumin levels | Baseline and 6 weeks

SECONDARY OUTCOMES:
Number of patients with adverse events | 8 weeks
  6 weeks of therapy and 2 weeks of follow-up post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Thadhani, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kalim S, Ortiz G, Trottier CA, Deferio JJ, Karumanchi SA, Thadhani RI, Berg AH. The Effects of Parenteral Amino Acid Therapy on Protein Carbamylation in Maintenance Hemodialysis Patients. J Ren Nutr. 2015 Jul;25(4):388-92. doi: 10.1053/j.jrn.2015.01.019. Epub 2015 Mar 5. PMID 25753604